CLINICAL TRIAL: NCT06211478
Title: Role of Vitamin E as an Adjuvant Therapy for Patients With Gaucher Disease Under Enzyme Replacement Therapy in Relation to Oxidative Stress
Brief Title: Role of Vitamin E in Gaucher Disease Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amira Abd el moneam, professor of pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD72/2022
Record Dates: First submitted 2024-01-09; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease | interventions — Vitamin E

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cases who are taking vitamin E (Experimental): gaucher disease patients with oxidative stress and vitamin E defeciency taking vitamin E treatment (weigh below 20 kg dose will be 200mg daily and whose weight above 20 kg dose will be 400mg daily for duration 6 months )
  Interventions: Drug: Vitamin E
- controls who are not taking vitamin E treatment (No Intervention): gaucher disease patients with oxidative stress and vitamin E defeciency not taking vitamin E treatment but take the standard of care which is enzyme replacement therapy

INTERVENTIONS:
Drug: Vitamin E — Vitamin E will be taken for 6 months for gaucher disease patients who have oxidative stress and vitamin E defecient
  Other Names: No other alternatives
  Arms: cases who are taking vitamin E

SUMMARY:
gaucher disease (GD) can be classified into three clinical types .type 1,the most common type ,is the chronic non neuronpathic form of the disease,which shows gighly variable signs and symptoms and variable course,with visceral,skeletal and hematologic involvement among others.the neurologocal involvement can be observed in types 2 and 3

DETAILED DESCRIPTION:
enzymatic defeciency in gaucher disease patients may induce a cascade of events that result in side effects, such as the production of reactive oxygen species(ROS) and reactive nitrogen species(RNS) that can then generate the oxidative stress whereas in body of healthy individuals,the production and degradation of ROS and RNS are generally balanced.

neurochemical abnormalities in patients with gaucher disease might be related to oxidative stress and inflammation in the brain.

oxidative stress induces peroxiredoxin-2 as cytoprotective response against RNS .it is able to detoxify a vast range of organic peroxides.

vitamin E well accepted nature most effective lipid soluble chain breaking antioxidant .

ELIGIBILITY:
Inclusion Criteria:

children and adolescents aged fron 2 to 18 years old with gaucher disease both type 1 and type 3 diagnosed clinically and confirmed by laboratory analysis patients who are on stable enzyme replacement therapy for at least 6 months -

Exclusion Criteria:

patients with infection or another inflammatory condition patients on multivitamin therapy known chronic liver disease (viral hepatitis,HIV) patients with renal impairement defined as creatinine level greater 1.2 for female and greater than 1.4 for male.

-

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — self representation of gender identity
Enrollment: 40 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
effect of vitamin E on oxidative stress and antioxidant markers in gaucher disease patients | 6 months
  Measuring the oxidative stress markers in gaucher disease MDA and anti oxidant markers which are peroxiredoxin 2 ,Glutathione peroxidase,superoxide dismutase and reduced glutathione

CONTACTS AND LOCATIONS:
Overall Officials: Amira A Adly, Phd, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pacheco N, Uribe A. Enzymatic analysis of biomarkers for the monitoring of Gaucher patients in Colombia. Gene. 2013 May 25;521(1):129-35. doi: 10.1016/j.gene.2013.03.044. Epub 2013 Mar 21. PMID 23523857
- [Background] Kartha RV, Terluk MR, Brown R, Travis A, Mishra UR, Rudser K, Lau H, Jarnes JR, Cloyd JC, Weinreb NJ. Patients with Gaucher disease display systemic oxidative stress dependent on therapy status. Mol Genet Metab Rep. 2020 Dec 9;25:100667. doi: 10.1016/j.ymgmr.2020.100667. eCollection 2020 Dec. PMID 33335836
- [Derived] Adly AAM, Ismail EAR, Ibrahim FA, Atef M, El Sayed KA, Aly NH. A 6-month randomized controlled trial for vitamin E supplementation in pediatric patients with Gaucher disease: Effect on oxidative stress, disease severity and hepatic complications. J Inherit Metab Dis. 2025 Jan;48(1):e12792. doi: 10.1002/jimd.12792. Epub 2024 Aug 25. PMID 39183538